CLINICAL TRIAL: NCT00960804
Title: A PHASE 3, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER, LONG-TERM SAFETY STUDY OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE OR HIP
Brief Title: Long-Term Study Of The Safety Of Tanezumab In Arthritis Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091040; NERVE FUNCTION EXTENSION STUDY (Other: Alias Study Number)
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tanezumab 5 mg (Experimental)
  Interventions: Biological: Tanezumab
- Tanezumab 10 mg (Experimental)
  Interventions: Biological: Tanezumab
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tanezumab — IV, 5 mg dose, q 8 weeks, for up to 80 weeks
  Arms: Tanezumab 5 mg
Biological: Tanezumab — IV, 10 mg dose, q 8 weeks, for up to 80 weeks
  Arms: Tanezumab 10 mg
Other: Placebo — IV, q 8 weeks, for up to 80 weeks
  Arms: Placebo

SUMMARY:
Tanezumab, administered for up to 1 1/2 years, reduces the pain of osteoarthritis without affecting how nerve impulses are transmitted in sensory nerves

DETAILED DESCRIPTION:
This study was terminated on 11 Nov 2010 following a US FDA clinical hold for tanezumab osteoarthritis clinical studies which halted dosing and enrollment of patients on 23 June 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Patients must consent in writing to participate in the study.
* Patients must be willing to comply with study visit schedule and study requirements, including, for women of child-bearing potential or male patients with female partners of child-bearing potential, the use of 2 forms of birth control, one of which is a barrier method.
* Patients must have participated in the A4091026 study.

Exclusion Criteria:

* Withdrawn from the A4091026 study for an adverse event or serious adverse event.
* Pregnant women, lactating mothers, women suspected of being pregnant, and women who wish to be pregnant during the course of clinical study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02-15 (Actual); Primary Completion 2010-11-11 (Actual); Study Completion 2010-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Jem Research, LLC, Atlantis, Florida
  - Medical Specialists of the Palm Beaches, Atlantis, Florida
  - Clinical Physiology Associates, Clinical Study Center, Fort Myers, Florida
  - Harris Bonnette, MD, Fort Myers, Florida
  - Arthritis & Rheumatic Care Center, South Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Neuroscience Consultants, LLC, South Miami, Florida
  - Asheville Imaging, Asheville, North Carolina
  - Biltmore Medical Associates, Asheville, North Carolina
  - Clinical Study Center of Asheville, LLC, Asheville, North Carolina
  - Asheville Neurology, Asheville, North Carolina
  - Ohio Research Center, Toledo, Ohio
  - Blair Neurologic Associates, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Coastal Carolina Research Center in Goose Creek, Goose Creek, South Carolina
  - Tidewater Neurology, Goose Creek, South Carolina
  - Neurodiagnostic Laboratories of San Antonio, Inc, San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091040&StudyName=Long-Term%20Study%20Of%20The%20Safety%20Of%20Tanezumab%20In%20Arthritis%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who received study drug and had end of study nerve function assessment data in previous study A4091026 (NCT00863772) were eligible to be enrolled in this study. Dosing interval between last dose in A4091026 (NCT00863772) and first dose in this study was not less than 8 weeks or more than 12 weeks.
Groups:
- Tanezumab 5 mg + Standard of Care: Participants who had previously received tanezumab (RN624 or PF-04383119) 5 milligram (mg) intravenous infusion in parent study A4091026 (NCT00863772), received tanezumab 5 mg intravenous infusion over 5 minutes every 8 weeks along with standard of care (SOC) as per investigator's discretion up to 32 weeks. SOC included analgesic medications (opioids, topical analgesics, non-steroidal anti-inflammatory drugs [NSAIDs], capsaicin products, injectable corticosteroids, and viscosupplementation) approved by United States Food and Drug Administration (FDA) or other applicable Health Authorities.
- Tanezumab 10 mg + Standard of Care: Participants who had previously received tanezumab (RN624 or PF-04383119) 10 mg intravenous infusion in parent study A4091026 (NCT00863772), received tanezumab 10 mg intravenous infusion over 5 minutes every 8 weeks along with SOC as per investigator's discretion up to 32 weeks. SOC included analgesic medications (opioids, topical analgesics, NSAIDs, capsaicin products, injectable corticosteroids, and viscosupplementation) approved by United States FDA or other applicable Health Authorities.
- Placebo + Standard of Care: Participants who had previously received placebo matched to tanezumab (RN624 or PF-04383119) intravenous infusion in parent study A4091026 (NCT00863772), received placebo matched to tanezumab intravenous infusion over 5 minutes every 8 weeks along with SOC as per investigator's discretion up to 32 weeks. SOC included analgesic medications (opioids, topical analgesics, NSAIDs, capsaicin products, injectable corticosteroids, and viscosupplementation) approved by United States FDA or other applicable Health Authorities.
Period: Overall Study
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Started | 7 | 4 | 10
Completed | 0 | 0 | 0
Not Completed | 7 | 4 | 10
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Study terminated by the sponsor | 5 | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care | Total
Number analyzed (Participants) | 7 | 4 | 10 | 21
Age, Customized [Count of Participants; unit: Participants]
  45 to 64 years | 7 | 2 | 6 | 15
  Greater than or equal to (>=) 65 years | 0 | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 10
  Male | 4 | 1 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From A4091026 (NCT00863772) Baseline in 5 Nerve Conduction Tests, Normal Deviate and Heart Rate-Deep Breathing, Normal Deviate (5NC [nd] + HRdb-[nd]) Composite Score at Week 24
Description: 5NC(nd)+HRdb(nd)composite score included 5 Nerve Conduction Studies(NCS)attributes(peroneal motor nerve distal latency [MNDL],peroneal nerve compound muscle action potential[CMAP],peroneal motor nerve conduction velocity[MNCV],tibial MNDL,sural sensory nerve action potential amplitude [SNAP])and HRdb value. Values of attributes scored as percentile(calculated from distribution of normal values corresponding to participant's baseline demographic characteristics),then expressed as normal deviate(nd)score based on standard normal distribution.Score >0=worse response,less than(<)0=better response compared to normal matched population.Score change>0=worsening,<0=improvement compared to baseline.2 neurological visits(NVs) were conducted both at baseline and Week 24. NCS measurements were collected once at each NV.HRdb measurements were collected twice and highest nd score was selected at each NV. Mean of selected measurements at each NV was calculated to obtain Baseline and Week 24 values.
Time Frame: A4091026: Baseline, A4091040: Week 24
Population: Intent-to-treat (ITT) analysis set included all participants who received at least 1 dose of intravenous study medication during this study A4091040. Missing values were imputed using last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
normal deviate score
  Baseline | 1.37 (3.19) | 2.96 (1.02) | 0.31 (2.76)
  Change at Week 24 | 0.28 (2.57) | 1.79 (2.70) | -1.40 (2.83)

2. Secondary Outcome: Change From A4091026 (NCT00863772) Baseline in Neuropathy Impairment Score- Lower Limb (NIS-LL) at Week 24
Description: NIS-LL:assess muscle weakness, reflexes, sensation;scored separately for left, right limbs. Components of muscle weakness (hip and knee flexion,hip and knee extension,ankle dorsiflexors,ankle plantar flexors,toe extensors,toe flexors) scored on scale 0(normal) to 4(paralysis),higher score=greater weakness. Components of reflexes(quadriceps femoris,triceps surae);sensation (touch pressure,pin-prick,vibration,joint position) scored 0=normal,1=decreased, or 2=absent. NIS-LL score: sum of scores of NIS items 17-24, 28-29 and 34-37. Total possible NIS-LL score range 0-88,high score=more impairment.
Time Frame: A4091026: Baseline, A4091040: Week 24
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication during this study A4091040. Missing values were imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Change at Week 24 | 1.14 (3.02) | 0.00 (0.00) | 0.00 (0.00)

3. Secondary Outcome: Change From A4091026 (NCT00863772) Baseline in Neuropathy Impairment Score (NIS) at Week 24
Description: NIS: 74 items, assess muscle weakness, reflexes and sensation; scored separately for left, right limbs (37 items for each side). Components of muscle weakness (hip and knee flexion, hip and knee extension, ankle dorsiflexors, ankle plantar flexors, toe extensors, toe flexors) scored on scale 0 (normal) to 4 (paralysis), higher score=greater weakness. Components of reflexes (quadriceps femoris, triceps surae) and sensation (touch pressure, pin-prick, vibration, joint position) scored 0 = normal, 1= decreased, or 2 = absent. Total possible NIS score range 0-244, higher score=greater impairment.
Time Frame: A4091026: Baseline, A4091040: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Change at Week 24 | 2.00 (5.29) | 0.00 (0.00) | 0.00 (0.00)

4. Secondary Outcome: Change From A4091026 (NCT00863772) Baseline in Neuropathy Symptoms and Change (NSC) Score at Week 24
Description: NSC score is the number of the 38 symptom questions where the participants indicated experiencing the symptom to any severity. Total score range: 0 to 38 where higher score indicated more symptoms.
Time Frame: A4091026: Baseline, A4091040: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
units on a scale
  Baseline | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Change at Week 24 | 0.00 (0.00) | 0.25 (0.50) | 0.10 (0.32)

5. Other Pre Specified Outcome: Change From A4091026 (NCT00863772) Baseline in 5 Nerve Conduction Tests, Normal Deviate (5NC [nd]) Score at Week 24
Description: 5NC (nd) score included five NCS attributes: peroneal MNDL, CMAP, MNCV; tibial MNDL; sural SNAP. Values of attributes scored as percentiles (calculated from distribution of normal values corresponding to participant's baseline demographic characteristics), then expressed as nd score based on standard normal distribution. For CMAP, MNCV, SNAP: score <0 indicated worse and >0 indicated better response; for peroneal,tibial MNDL: score >0 indicated worse and <0 indicated better response, as compared to normal matched population. For CMAP, MNCV, SNAP: score change <0 indicated worsening and >0 indicated improvement; for peroneal,tibial MNDL: score change >0 indicated worsening and <0 indicated improvement, as compared to baseline. Total score calculated as sum of each NCS attribute. Total score >0 indicated worse and <0 indicated better response as compared to normal matched population. Total score change >0 indicated worsening and <0 indicated improvement as compared to baseline.
Time Frame: A4091026: Baseline, A4091040: Week 24
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication during this study A4091040. Missing values were imputed using LOCF method. 'Number Analyzed' signifies participants evaluated at specific time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
normal deviate score
  Baseline: Peroneal CMAP | -0.20 (1.16) | -0.85 (0.45) | 0.13 (1.27)
  Baseline: Peroneal MNCV | 0.61 (1.55) | 1.03 (1.02) | 0.77 (1.78)
  Baseline: Peroneal MNDL | -0.14 (0.70) | 0.33 (0.51) | -0.09 (0.93)
  Baseline: Tibial MNDL | 0.82 (1.24) | 1.41 (1.12) | 0.97 (0.61)
  Baseline: Sural SNAP | -0.95 (0.95) | -0.80 (1.04) | -0.72 (1.14)
  Baseline: 5NC (nd) composite score | 1.21 (2.90) | 2.37 (1.38) | 0.69 (2.71)
  Change at Week 24: Peroneal CMAP: number analyzed (Participants) | 7 | 3 | 9
  Change at Week 24: Peroneal CMAP | -1.03 (1.33) | -0.32 (0.45) | -0.02 (0.75)
  Change at Week 24: Peroneal MNCV: number analyzed (Participants) | 7 | 2 | 9
  Change at Week 24: Peroneal MNCV | -0.16 (0.81) | -0.50 (0.40) | 0.16 (1.19)
  Change at Week 24: Peroneal MNDL: number analyzed (Participants) | 7 | 2 | 9
  Change at Week 24: Peroneal MNDL | -0.06 (1.34) | -0.82 (0.40) | -0.08 (0.71)
  Change at Week 24: Tibial MNDL: number analyzed (Participants) | 7 | 3 | 9
  Change at Week 24: Tibial MNDL | -0.89 (1.42) | -0.38 (0.39) | -0.59 (1.15)
  Change at Week 24: Sural SNAP: number analyzed (Participants) | 7 | 3 | 9
  Change at Week 24: Sural SNAP | -0.29 (0.78) | -0.49 (0.57) | 0.14 (1.01)
  Change at Week 24:5NC(nd) composite score: number analyzed (Participants) | 7 | 3 | 9
  Change at Week 24:5NC(nd) composite score | 0.53 (2.21) | 1.33 (2.96) | -0.96 (2.40)

6. Other Pre Specified Outcome: Change From A4091026 (NCT00863772) Baseline in Heart Rate-Deep Breathing, Normal Deviate (HRdb, [nd]) Score at Week 24
Description: HRdb test was used to evaluate the effect of treatment on autonomic function. Participant took a series of 8 deep breaths and average heart rate difference was measured and compared to normative data. R-R (time between two consecutive R waves in the electrocardiogram) response to deep breathing was reported as normal deviates. Score <0 indicated worse response and >0 indicated better response as compared to normal matched population. Score change <0 indicated worsening and >0 indicated improvement as compared to baseline. 2 neurological visits (NVs) were conducted both at baseline and Week 24. Measurements were collected twice and highest nd score was selected at each NV. Mean of the selected measurements was calculated to obtain Baseline and Week 24 values.
Time Frame: A4091026: Baseline, A4091040: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: normal deviate score
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
normal deviate score
  Baseline | -0.16 (0.59) | -0.59 (0.36) | 0.38 (1.15)
  Change at Week 24 | 0.25 (0.53) | -0.17 (0.35) | -0.21 (0.54)

7. Other Pre Specified Outcome: Change From A4091026 (NCT00863772) Baseline in Intraepidermal Nerve Fiber Density (IENF) at Week 24
Description: IENF density was quantified in 3 millimeter (mm) immunostained (PGP 9.5 immunohistochemical staining) skin punch biopsies taken from the distal end of the leg, 10 centimeter (cm) above the lateral malleolus, within the territory of the sural nerve, containing epidermis and superficial dermis to evaluate amount of small diameter nerve fibers. Skin biopsies were taken from normal appearing skin and skin having local scar, signs of trauma, ulceration, or active dermatologic process were avoided.
Time Frame: A4091026: Baseline, A4091040: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nerve fiber count/millimeter
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
nerve fiber count/millimeter
  Baseline | 13.01 (6.54) | 8.99 (5.79) | 9.75 (4.46)
  Change at Week 24 | -0.90 (3.02) | 0.07 (1.47) | 0.67 (4.26)

8. Other Pre Specified Outcome: Change From A4091026 (NCT00863772) Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Domain Scores at Week 8, 16, 24 and 32
Description: WOMAC Index: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items), and physical function (17 items) in participants with osteoarthritis of the index hip or index knee. Each question was assessed on Numeric Rating Scale (NRS) as 0(none) to 10(extreme).Total possible domain score was calculated as the mean of the score for each domain questions. Score range:0-10,high scores=high pain/stiffness/difficulty in physical activity.
Time Frame: A4091026: Baseline, A4091040: Week 8, 16, 24, 32
Population: ITT analysis set included all participants who received at least 1 dose of intravenous study medication during this study A4091040. Missing values were imputed using LOCF method. Results were not reported at Week 32 as none of the participants were evaluable for this measure at Week 32.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
units on a scale
  Baseline: Pain | 5.66 (2.03) | 6.75 (1.04) | 6.70 (1.85)
  Baseline: Physical Function | 6.01 (1.50) | 6.88 (0.92) | 6.73 (1.94)
  Baseline: Stiffness | 6.64 (1.97) | 6.88 (0.25) | 6.65 (2.00)
  Change at Week 8: Pain | -3.20 (2.61) | -4.45 (3.23) | -2.76 (2.03)
  Change at Week 8: Physical Function | -3.38 (2.50) | -4.60 (2.88) | -2.24 (1.78)
  Change at Week 8: Stiffness | -3.86 (3.01) | -4.75 (2.96) | -2.25 (2.84)
  Change at Week 16: Pain | -2.91 (2.66) | -5.05 (2.04) | -2.84 (2.00)
  Change at Week 16: Physical Function | -3.26 (2.46) | -5.22 (1.66) | -2.42 (2.04)
  Change at Week 16: Stiffness | -3.79 (2.91) | -5.25 (2.02) | -2.50 (2.89)
  Change at Week 24: Pain | -2.91 (2.66) | -5.05 (2.04) | -2.82 (2.00)
  Change at Week 24: Physical Function | -3.26 (2.46) | -5.22 (1.66) | -2.42 (2.03)
  Change at Week 24: Stiffness | -3.79 (2.91) | -5.25 (2.02) | -2.50 (2.89)

9. Other Pre Specified Outcome: Change From A4091026 (NCT00863772) Baseline in Patient's Global Assessment (PGA) of Osteoarthritis at Week 8, 16, 24 and 32
Description: PGA: Participants answered the following question: "Considering all the ways your osteoarthritis in your knee or hip affects you, how are you doing today?" Participants rated their condition using a 5-point Likert scale. Score range: 1 to 5. 1: Very Good (asymptomatic and no limitation of normal activities); 2: Good (mild symptoms and no limitation of normal activities); 3: Fair (moderate symptoms and limitation of some normal activites); 4: Poor (severe symptoms and inability to carry out most normal activities); 5: Very Poor (very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: A4091026: Baseline, A4091040: Week 8, 16, 24, 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
units on a scale
  Baseline | 3.00 (0.00) | 3.50 (0.58) | 3.70 (0.82)
  Change at Week 8 | -0.86 (1.07) | -2.00 (0.00) | -1.10 (1.10)
  Change at Week 16 | -1.00 (1.00) | -2.00 (0.00) | -1.20 (0.92)
  Change at Week 24 | -1.00 (1.00) | -2.00 (0.00) | -1.30 (0.82)

10. Other Pre Specified Outcome: Percentage of Participants With Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Response
Description: OMERACT-OARSI response: >=50 percent (%) improvement from A4091026 (NCT00863772) baseline and absolute change from A4091026 (NCT00863772) baseline of >=2 units at week of interest in WOMAC pain or physical function subscales, or at least 2 of the following 3 being true: >=20% improvement from A4091026 (NCT00863772) baseline and absolute change from A4091026 (NCT00863772) baseline of >=1 unit at week of interest in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis (score: 1-5, higher score=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score: 0-10, higher score=higher pain/difficulty).
Time Frame: Week 8, 16, 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
percentage of participants
  Week 8 | 85.7 | 75.0 | 70.0
  Week 16 | 85.7 | 100.0 | 70.0
  Week 24 | 85.7 | 100.0 | 70.0

11. Other Pre Specified Outcome: Change From A4091026 (NCT00863772) Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 8, 16 and 24
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items) and physical function (17 items) in participants with osteoarthritis of knee or hip. WOMAC average score is the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 to 10, where higher score indicates worse response. Change from baseline <0 indicates an improvement.
Time Frame: A4091026: Baseline, A4091040: Week 8, 16, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
units on a scale
  Baseline | 6.10 (1.71) | 6.83 (0.67) | 6.69 (1.88)
  Change at Week 8 | -3.48 (2.58) | -4.60 (2.99) | -2.42 (2.15)
  Change at Week 16 | -3.32 (2.56) | -5.17 (1.85) | -2.59 (2.23)
  Change at Week 24 | -3.32 (2.56) | -5.17 (1.85) | -2.58 (2.23)

12. Other Pre Specified Outcome: Percentage of Participants With at Least 30%, 50%, 70% and 90% Reduction From A4091026 (NCT00863772) Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint (knee or hip) during the past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicate higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicate higher pain.
Time Frame: Week 8, 16, 24, 32
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
percentage of participants
  Week 8: >=30% Reduction | 85.7 | 75.0 | 60.0
  Week 8: >=50% Reduction | 42.9 | 75.0 | 60.0
  Week 8: >=70% Reduction | 42.9 | 75.0 | 10.0
  Week 8: >=90% Reduction | 14.3 | 50.0 | 10.0
  Week 16: >=30% Reduction | 71.4 | 75.0 | 60.0
  Week 16: >=50% Reduction | 42.9 | 75.0 | 60.0
  Week 16: >=70% Reduction | 42.9 | 75.0 | 20.0
  Week 16: >=90% Reduction | 14.3 | 50.0 | 10.0
  Week 24: >=30% Reduction | 71.4 | 75.0 | 60.0
  Week 24: >=50% Reduction | 42.9 | 75.0 | 60.0
  Week 24: >=70% Reduction | 42.9 | 75.0 | 20.0
  Week 24: >=90% Reduction | 14.3 | 50.0 | 10.0
  Week 32: >=30% Reduction | 71.4 | 75.0 | 60.0
  Week 32: >=50% Reduction | 42.9 | 75.0 | 60.0
  Week 32: >=70% Reduction | 42.9 | 75.0 | 20.0
  Week 32: >=90% Reduction | 14.3 | 50.0 | 10.0

13. Other Pre Specified Outcome: Percentage of Participants With Improvement of At Least 2 Points From A4091026 (NCT00863772) Baseline in Patient's Global Assessment (PGA) of Osteoarthritis
Description: as for outcome 9
Time Frame: Week 8, 16, 24, 32
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
percentage of participants
  Week 8 | 0 | 0 | 10.0
  Week 16 | 0 | 0 | 10.0
  Week 24 | 0 | 0 | 20.0
  Week 32 | 0 | 0 | 20.0

14. Other Pre Specified Outcome: Change From A4091026 (NCT00863772) Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Domain Scores at Week 24
Description: SF-36v2 is a self-administered questionnaire evaluating 8 aspects/domains of functional health and wellbeing: physical function, role physical, bodily pain, vitality, general health, social function, role emotional and mental health. The total score for each domain is scaled 0-100 (100 = highest level of functioning). Change from baseline >0 indicates an improvement.
Time Frame: A4091026: Baseline, A4091040: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
units on a scale
  Baseline: General Health | 67.71 (16.18) | 79.50 (9.57) | 77.40 (9.61)
  Baseline: Physical Function | 55.00 (24.15) | 47.50 (35.24) | 39.00 (23.43)
  Baseline: Role Physical | 66.96 (23.31) | 53.13 (36.98) | 34.38 (26.88)
  Baseline: Bodily Pain | 51.14 (25.20) | 42.25 (22.54) | 33.50 (19.05)
  Baseline: Vitality | 54.46 (21.56) | 59.38 (15.73) | 61.88 (24.02)
  Baseline: Social Function | 82.14 (20.23) | 78.13 (25.77) | 82.50 (17.87)
  Baseline: Role Emotional | 79.76 (20.33) | 79.17 (25.00) | 70.83 (21.61)
  Baseline: Mental Health | 73.57 (16.26) | 81.25 (8.54) | 87.00 (14.38)
  Change at Week 24: General Health | 1.57 (12.22) | 6.25 (4.79) | -3.90 (13.10)
  Change at Week 24: Physical Function | 14.29 (27.60) | 25.00 (10.80) | 5.00 (32.32)
  Change at Week 24: Role Physical | 8.04 (25.95) | 31.25 (24.47) | 17.50 (14.37)
  Change at Week 24: Bodily Pain | 8.00 (35.23) | 34.75 (14.03) | 13.60 (19.39)
  Change at Week 24: Vitality | 7.14 (14.17) | 17.19 (11.83) | 3.75 (5.27)
  Change at Week 24: Social Function | 3.57 (11.89) | 21.88 (25.77) | 0.00 (15.59)
  Change at Week 24: Role Emotional | -2.38 (30.32) | 6.25 (29.95) | 5.00 (23.31)
  Change at Week 24: Mental Health | 1.43 (14.06) | 8.75 (8.54) | -5.50 (8.32)

15. Other Pre Specified Outcome: Change From A4091026 (NCT00863772) Baseline in 36-Item Short-Form Health Survey Version 2 (SF-36v2) Physical and Mental Component Scores at Week 24
Description: SF-36v2 is a self-administered questionnaire evaluating 8 aspects/domains of functional health and wellbeing: physical function, role physical, bodily pain, vitality, general health, social function, role emotional and mental health. Total score for each aspect were scaled 0-100 (100=highest level of functioning). For obtaining physical and mental component scores, z-score for each scale = (observed score -mean score for general 1990 United States [US] population)/corresponding standard deviation. The 2 component scores were obtained by multiplying each aspect z-score by physical or mental factor score coefficient (1990 general US population) and summing the eight products. Component scores indicated how many standard deviations higher (in case of positive z-score [better functioning])/lower (in case of negative z-score [worse functioning]) participant's value was relative to the mean of the reference population. Change from baseline >0 indicates an improvement.
Time Frame: A4091026: Baseline, A4091040: Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Number analyzed (Participants) | 7 | 4 | 10
z-score
  Baseline: Mental Component Score | 0.17 (0.92) | 0.55 (0.61) | 0.83 (1.17)
  Baseline: Physical Component Score | -0.95 (1.08) | -1.33 (1.04) | -1.88 (0.63)
  Change at Week 24: Mental Component Score | -0.09 (0.90) | 0.28 (0.93) | -0.19 (0.50)
  Change at Week 24: Physical Component Score | 0.50 (1.03) | 1.27 (0.39) | 0.50 (0.95)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tanezumab 5 mg + Standard of Care | Tanezumab 10 mg + Standard of Care | Placebo + Standard of Care
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/4 | 0/10
Other Adverse Events (participants affected / at risk) | 6/7 | 3/4 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 5 mg + Standard of Care (N=7) | Tanezumab 10 mg + Standard of Care (N=4) | Placebo + Standard of Care (N=10)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 5 mg + Standard of Care (N=7) | Tanezumab 10 mg + Standard of Care (N=4) | Placebo + Standard of Care (N=10)
Vitreous floaters (Eye disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Nerve conduction studies abnormal (Investigations) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to FDA-imposed clinical hold, enrollment stopped prematurely, thus inadequate power to fulfill primary objectives.Efficacy data beyond Week 32 not collected.Change in planned analysis added results of >=70%, 90% reduction in WOMAC pain subscale.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.